CLINICAL TRIAL: NCT03312361
Title: Assessing Air Travel Safety in Neuromuscular Dystrophy: Standard Versus Prolonged High Altitude Simulation Tests
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Reshma Amin, Respirologist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1000051539
Record Dates: First submitted 2017-10-12; First posted 2017-10-17 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Neuromuscular Diseases; High Altitude Hypoxia
MeSH Terms: conditions — Neuromuscular Diseases | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 15% Oxygen (Experimental): All participants will breath in 15% oxygen for 2 hours
  Interventions: Drug: 15% oxygen

INTERVENTIONS:
Drug: 15% oxygen — Participants will inhale 15% oxygen for 2 hours to see how it affects them.

SUMMARY:
To determine if a prolonged high altitude simulation test (HAST) lasting two hours, identifies more patients at risk of respiratory failure than the standard HAST lasting 20 minutes, in patients with neuromuscular disease (NMD) and severe pulmonary restriction. To evaluate the safety of supplemental oxygen administered in those with a positive HAST in the NMD population.

DETAILED DESCRIPTION:
Study Procedures

Patients were screened for eligibility during a regularly scheduled clinic visit in which spirometry was performed in accordance with the American Thoracic Society recommendations.4 If eligible, they were approached by a Research Coordinator and invited to participate in the study. The study visit was organized within 4 weeks of screening and included both diagnostic and (if applicable) therapeutic HCT trials. After enrolment, patients' local medical records were reviewed for baseline data.

Baseline Assessment:

On the day of the HCT, a brief focused history including current respiratory symptoms was performed. Study participants sat for a minimum of 5 minutes before baseline measurements were taken. Vital signs (heart rate, respiratory rate, blood pressure), capillary blood gas, transcutaneous capnography and pulse oximetry were performed immediately prior to the start of testing. The transcutaneous CO2 and SpO2 values obtained just prior to provision of the gas mixture were considered the baseline values.

Testing Procedures: Study participants underwent a standard 20 minute HCT and if eligible (i.e. not positive or test not terminated) then immediately continued on to complete the 120 minute extended HCT. A gas mixture of 15% oxygen in nitrogen from a specially prepared cylinder was administered via a non-rebreather mask sealed to the face. Flow was adjusted for patient comfort, and to match inspiratory flow by maintaining non-rebreather bag inflation thus ensuring no entrainment of room air (between 6-15 L/minute). The patient would breathe this mixture for up to 120 minutes, or until they met stopping criteria. Continuous pulse oximetry, transcutaneous capnography and respiratory rate were recorded throughout the HCT. Patients were asked to indicate the severity of dyspnea every 10 minutes using the modified Borg scale. Capillary blood gases were drawn at the end of the standard and prolonged HCTs (i.e. immediately after 20 and 120 minutes, respectively). The patient was observed for 20 minutes after completion of the HCT, or until oxygen saturation and transcutaneous pCO2 returned to baseline levels. The HCT was considered positive and the test was stopped if any of the following occurred: i) oxygen saturation <88% for two consecutive minutes (as per institutional cutoff for prescription of oxygen); ii) ≥ 10mmHg rise from baseline in transcutaneous CO2 sustained for 2 minutes and confirmed by capillary blood gas; iii) severe symptoms such as dyspnea or confusion; iv) or participant request to stop testing. Repeat complete vital signs were performed prior to the end of the study visit.

ELIGIBILITY:
Inclusion Criteria:

* individuals with a confirmed diagnosis of NMD
* age ≥ 5 years of age
* absence of hypoxia at rest, defined as oxygen saturation ≥ 92% for two consecutive minutes while at rest and breathing room air
* absence of daytime hypercapnea at rest, defined by partial pressure of carbon dioxide (pCO2) less than 45 mmHg on capillary or arterial blood gas at rest
* patient or authorized substitute decision maker provides consent to study participation.

Exclusion Criteria:

* current respiratory tract infection
* inability to comply with the study procedures
* severe heart failure as defined by uncontrolled symptoms of heart failure, or left ventricular ejection fraction < 30%
* presence of a tracheostomy
* use of domiciliary bilevel positive airway pressure (BPAP) for more than 12 hours daily
* recent hospital admission within the past 4 weeks.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Prolonged high altitude simulation test | 3 years
  To determine if a prolonged high altitude simulation test (HAST) lasting two hours, identifies more patients at risk of respiratory failure than the standard HAST lasting 20 minutes, in patients with NMD and severe pulmonary restriction

SECONDARY OUTCOMES:
Interventional high altitude simulation test | 3 years
  In patients with a positive standard or prolonged HAST, we will evaluate the safety of supplemental oxygen administered during a HAST for this population

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No